CLINICAL TRIAL: NCT00223015
Title: Investigation of the Steady State Pharmacokinetics of Tacrolimus, Mycophenolate Mofetil and Fluvastatin After Renal Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 002
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2005-10-20 (Estimated); Status verified 2004-05

CONDITIONS: Renal Transplantation
Keywords: renal transplantation; pharmacokinetics; Fluvastatin; Mycophenolat mofetil; tacrolimus
MeSH Terms: interventions — Fluvastatin; Tacrolimus

INTERVENTIONS:
Drug: Fluvastatin, Tacrolimus, Mycophenolat Mofetil

SUMMARY:
Steady state pharmacokinetics of tacrolimus, mycophenolat mofetil and fluvastatin in renal transplant patients are investigated to look for potential interaction between these drugs.

All patient enrolled in this PKI-Study had no changes in the therapy before or because of the study. Only patients without changes more than 4 weeks were included

ELIGIBILITY:
Inclusion Criteria:

* renal transplant patients (18 - 65 years, inclusive)
* cadaver and living renal transplants(1. Ntx, 2. Ntx)
* Immunsuppression: Tacrolimus with or without Mycophenolat Mofetil und and fluvastatin Fluvastatin for a minimum of three months
* writen informt consent by the patient

Exclusion Criteria:

* contraindications for statins
* pregnancy or lactating
* elevated liver or muscle encymes (> 2x up to normal values: AST, ALT, bilirubine, CPK)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2004-05; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Renders, MD, Principal Investigator — University of Schleswig-Holstein, campus Kiel Department odf Nephrology